CLINICAL TRIAL: NCT02923986
Title: A Phase Ib/IIa Single-arm, Open-label Clinical Trial to Evaluate the Safety, Pharmacokinetics, and Efficacy of BP1001 (a Liposomal Grb2 Antisense Oligonucleotide) in Combination With Dasatinib in Patients With Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia (CML) Including Chronic Phase Patients Who Have Failed Initial Tyrosine Kinase Inhibitor (TKI) Therapy, Accelerated or Blast Phase, Ph+ Acute Myeloid Leukemia (AML) or High-risk Ph+ Myelodysplastic Syndrome (MDS)
Brief Title: Clinical Trial of BP1001 (Liposomal Grb2 Antisense Oligonucleotide) in Combination With Dasatinib in Patients With Ph + CML Who Have Failed TKI, Ph+ AML, Ph+ MDS
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No enrollment
Sponsor: Bio-Path Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP1001-202-CML
Record Dates: First submitted 2016-09-12; First posted 2016-10-05 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Chronic Myelogenous Leukemia, Ph1-Positive; Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: Liposomal Grb-2 treatment of Ph+ CML; Liposomal Grb-2 with Das for Ph+ CML; Liposomal Grb-2 treatment of Ph+ AML; Liposomal Grb-2 with Das for Ph+ AML; Liposomal Grb-2 treatment of Ph+ MDS; Liposomal Grb-2 with Das for Ph+ MDS
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Dasatinib; amsonic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BP1001 (varying dose) + Dasatinib (Experimental): Phase 1b: BP1001 (varying dose levels) in combination with Das
  Interventions: Drug: BP1001 (varying dose); Drug: Dasatinib
- BP1001 (fixed dose) + Dasatinib (Experimental): Phase IIa: BP1001 (fixed dose based on Phase 1b) in combination with Das
  Interventions: Drug: BP1001 (fixed dose); Drug: Dasatinib

INTERVENTIONS:
Drug: BP1001 (varying dose) — BP1001 (varying dose)
  Other Names: Liposomal Grb-2; L-Grb-2
  Arms: BP1001 (varying dose) + Dasatinib
Drug: BP1001 (fixed dose) — BP1001 (fixed dose)
  Other Names: Liposomal Grb-2; L-Grb-2
  Arms: BP1001 (fixed dose) + Dasatinib
Drug: Dasatinib — Dasatinib
  Other Names: Das

SUMMARY:
The primary objective of the Phase Ib study is to determine the dose-limiting toxicity (DLT) and maximal tolerated dose (MTD) of BP1001 in combination with dasatinib in patients with with Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia (CML) including chronic phase patients who have failed initial tyrosine kinase inhibitor (TKI) therapy, accelerated or blast phase, Ph+ Acute Myeloid Leukemia (AML) or High-risk Ph+ Myelodysplastic Syndrome (MDS). The primary objective of the Phase IIa study is to assess the efficacy of the combination of BP1001 and dasatinib in patients with Ph+ CML, Ph+AML, or high-risk Ph+ MDS.

DETAILED DESCRIPTION:
The Grb2 gene has been mapped to the human chromosome region 17q22-qter, a region that is duplicated in leukemias and solid tumors, which may result in an increased copy number of the Grb2 gene product. As Grb2 is important for the transformation of murine hematopoietic cells, and the proliferation of human leukemia cells that express high levels of oncogenic tyrosine kinases, inhibition of Grb2 may have a significant impact on the natural history of leukemias. The study drug (BP1001) may be able to inhibit the cells from making Grb-2. Researchers hope that without this protein, the leukemia cells will die.

Researchers hope that the combination of BP1001 and Das will provide a benefit to Ph+ CML patients, including chronic phase patients who have failed initial TKI therapy, accelerated or blast phase Ph+ AML, and high-risk Ph+ MDS patients.

This is a Phase Ib/IIa, multicenter, study of BP1001 in combination with Das in participants with Ph+ CML, including chronic phase patients who have failed initial TKI therapy, accelerated or blast phase Ph+ AML, and high-risk Ph+ MDS.

This is a Phase Ib/IIa, multicenter, study of BP1001 in combination with dasatinib in participants with Ph+ CML who are in chronic phase who have failed initial TKI therapy, accelerated or blast phase, Ph+ AML or high-risk Ph+ MDS.

This trial will utilize a single arm, open label design to assess the safety profile, DLT, MTD, PK, and efficacy of BP1001 in combination with dasatinib.

The Phase Ib study employs an open-label, sequential, dose-escalation design to assess safety, tolerability and toxicity, tumor response and anti-leukemic activity.

A standard "3+3" design will be used in which successive cohorts of patients are being treated with BP1001 at the MTD (or highest tested dose [HTD] if the MTD is not defined) and 1 level below the MTD (or HTD) in combination with a fixed dose of dasatinib to characterize safety and biological effect, as well as identify the recommended Phase IIa dose.

Up to 6 evaluable participants are expected to participate in the Phase Ib part of the study and up to 40 evaluable participants are expected to participate in the Phase IIa part of the study.

ELIGIBILITY:
Inclusion Criteria

At the time of Screening, participants must meet all of the following criteria to be considered eligible to participate in the study:

1. Adults ≥18 years of age
2. Females must be of non-childbearing potential, surgically sterile, postmenopausal, or practice adequate methods of contraception during the study and for 30 days after the last dose of study drug or dasatinib
3. Males must agree to use an adequate method of contraception during the study and for at least 30 days after the last dose of study drug or dasatinib
4. Histologically documented diagnosis of Ph+ CML including chronic phase patients who have failed initial TKI therapy, accelerated or blast phase, Ph+ AML or High-risk Ph+ MDS.

   Ph+ chronic phase CML patients who are resistant to 1 or more TKIs, including dasatinib. Dasatinib-resistant patients can enroll in the Phase Ib portion of the study but are excluded from the Phase IIa portion of the study.

   One of the following parameters is required to meet criteria for accelerated CML:
   * Blasts in Peripheral Blood or Bone Marrow ≥15%
   * Promyelocytes and Blasts in Peripheral Blood or Bone Marrow ≥30%
   * PB or BM basophils ≥20%
   * Thrombocytopenia <100 x 103/ml, not resulting from therapy
   * Cytogenetic clonal evolution CML blast phase is defined as ≥30% blasts in peripheral blood or bone marrow, or presence of extramedullary disease, except for liver or spleen.

   AML/MDS

   Ph+ AML is defined as:

   • Ph+ and meets diagnostic criteria for AML

   o Myeloid blasts ≥20 % or presence of AML-defining recurrent cytogenetic abnormality.

   Ph+ high-risk MDS defined as:

   • Ph+ high risk MDS ≥10% myeloid blasts or IPSS ≥intermediate-2
5. Adequate hepatic and renal functions as defined by:

   1. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 times the upper limit of normal (ULN); and
   2. Total bilirubin ≤1.5 times ULN; and
   3. Estimated glomerular filtration rate (eGFR) of at least 40 ml/min. These estimations can be calculated using any of the following methods (Appendix D):

   i. Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi) equation
   * GFR = 141 × min (Scr /κ, 1)α × max(Scr /κ, 1)-1.209 × 0.993Age × 1.018 [if female] × 1.159 [if black] ii. Cockcroft gault equation
   * Cockcroft Gault equation utilizing the TBW (Total body weight) to calculate an estimated creatinine clearance iii. CrCl = [(140 - age) x TBW] / (Scr x 72) x 0.85 [if female]
   * Modification of Diet in Renal Disease (MDRD) Study equation iv. GFR (mL/min/1.73 m2) = 175 × (Scr)-1.154 × (Age)-0.203 × 0.74 [if female] x 1.212 [if African American (AA)]
   * Creatinine clearance estimated by 24-hr urine collection for creatinine clearance
6. Documented Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
7. Recovered from the effects of any prior surgery, radiotherapy, or antineoplastic treatment (with the exception of alopecia), based on Investigator assessment
8. Willing and able to provide written informed consent

Exclusion Criteria

At the time of Screening, participants who meet any of the following criteria will be excluded from participating in the study:

1. Patients with T315I mutation will not be excluded, but their response will be analyzed separately.
2. Another primary malignancy other than CML, AML, or MDS within the past 2 years except non-melanoma skin cancer, or carcinoma in situ of the cervix.
3. Known, active leptomeningeal leukemia requiring intrathecal therapy. NOTE: Patients with a history of CNS disease may be allowed to participate based on at least 2 consecutive documented, negative spinal fluid assessment prior to Screening
4. Isolated extramedullary leukemia without also meeting bone marrow criteria for acute leukemia (i.e., ≥20% blasts in bone marrow aspirate)
5. Receipt of any anti-cancer therapy within 14 days of starting BP1001, with the exception of hydroxyurea or anagrelide, or TKI (within 2 days)
6. Uncontrolled active, untreated, or progressive infection
7. Receipt of any investigational agent within 14 days or 5 half-lives of starting BP1001
8. Females who are pregnant, test positive for pregnancy, or are breast-feeding during the Screening period, or intend to become pregnant or breast-feed during the course of the study or within 30 days after last dose of study drug
9. Prior exposure to BP1001
10. Patients with a history of intolerance to dasatinib or for whom dasatinib may not be appropriate
11. Serious intercurrent medical or psychiatric illness which, in the opinion of the Investigator, would interfere with the ability of the participant to complete the study
12. Known active or clinically significant hepatitis B infection (based on positive surface antigen [HBsAg]), hepatitis C infection (based on positive antibody [HCV Ab]), or human immunodeficiency virus (HIV-1 or HIV-2, based on positive antibody)
13. Presence of concurrent conditions that, in the opinion of the Investigator and/or Medical Monitor, may compromise the participant's ability to tolerate study treatment or interfere with any aspect of study conduct or interpretation of results. This includes but is not limited to, unstable or uncontrolled angina, New York Heart Association (NYHA) class III or IV congestive heart failure, uncontrolled and sustained hypertension, clinically significant cardiac dysrhythmia or clinically significant ECG abnormality (e.g., QTcF >470 msec)
14. Has had any of the following: clinically significant pleural effusion within 2 months, myocardial infarction, unstable angina pectoris, coronary/peripheral artery bypass graft, cerebrovascular accident or transient ischemic attack within 6 months.
15. Uncontrolled seizure disorder (i.e., seizures within the past 2 months).
16. Unable or unwilling to communicate or cooperate with the Investigator or follow the protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity of BP1001 using non-hematologic and hematologic parameters per NCI CTCAE criteria | 240 days
  Phase 1b portion of the study: Determine the dose limiting toxicity of BP1001 in combination with Das
Maximum Tolerated Dose of BP1001 using non-hematologic and hematologic parameters per NCI CTCAE criteria | 240 days
  Phase 1b portion of the study: Determine the maximum tolerated dose of BP1001 in combination with Das
Efficacy of the combination of BP1001 and Das using hematologic response by bone marrow aspirate or biopsy and complete blood counts | 240 days
  Phase IIa portion of the study: Assess the efficacy of the combination of BP1001 and Das
Efficacy of the combination of BP1001 and Das using cytogenetic response (karyotyping) by bone marrow aspirate or biopsy | 240 days
  Phase IIa portion of the study: Assess the efficacy of the combination of BP1001 and Das
Efficacy of the combination of BP1001 and Das using molecular response (PCR) by bone marrow aspirate or biopsy | 240 days
  Phase IIa portion of the study: Assess the efficacy of the combination of BP1001 and Das

SECONDARY OUTCOMES:
Safety of BP1001 in combination with Das using non-hematologic and hematologic parameters per NCI CTCAE criteria | 30 days
  Evaluate Safety of BP1001 in combination with Das
Efficacy of the combination of BP1001 and Das using hematologic response by bone marrow aspirate or biopsy and complete blood counts versus Das alone by historical outcome comparison | 240 days
  Determine whether the combination of BP1001 and Das provides greater efficacy (Hematologic Response) than Das alone (by historical comparison)
Efficacy of the combination of BP1001 and Das using cytogenetic response (karyotyping) by bone marrow aspirate or biopsy versus Das alone by historical outcome comparison | 240 days
  Determine whether the combination of BP1001 and Das provides greater efficacy (Cytogenetic Response) than Das alone (by historical comparison)
Efficacy of the combination of BP1001 and Das using molecular response (PCR) by bone marrow aspirate or biopsy versus Das alone by historical outcome comparison | 240 days
  Determine whether the combination of BP1001 and Das provides greater efficacy (Molecular Response) than Das alone (by historical comparison)
In vivo PK using plasma to compute half life and elimination | 30 days
  Evaluate in vivo PK of BP1001 when given alone and in combination with Das
Time to Response using hematologic response using bone marrow biopsy or aspirate and complete blood counts | 30 days
  Assess time to response from administration of BP1001 + Das to hematologic response
Time to Response using cytogenetic response (karyotyping) using bone marrow biopsy or aspirate | 30 days
  Assess time to response from administration of BP1001 + Das to cytogenetic response
Time to Response using molecular response (PCR) using bone marrow biopsy or aspirate | 30 days
  Assess time to response from administration of BP1001 + Das to molecular response
Duration of Response using hematologic response using bone marrow biopsy or aspirate and complete blood counts from day of response to day of disease progression | 30 days
  Assess duration of response from day of response to day of disease progression
Duration of Response using cytogenetic response (karyotyping) using bone marrow biopsy or aspirate from day of response to day of disease progression | 30 days
  Assess duration of response from day of response to day of disease progression
Duration of Response using molecular response (PCR) using bone marrow biopsy or aspirate from day of response to day of disease progression | 30 days
  Assess duration of response from day of response to day of disease progression
Overall Survival from date of study entry to study closure | 240 days
  Assess overall survival from date of study entry to study closure

CONTACTS AND LOCATIONS:
Overall Officials: Maro Ohanian, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No